CLINICAL TRIAL: NCT04158128
Title: The Clinical Implications and Functional Roles of Immune Checkpoint Pathways in Primary Central Nervous System Lymphomas
Brief Title: The Clinical Implications of Immune Checkpoint Pathways in PCNSL
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201608069RINB
Record Dates: First submitted 2019-02-15; First posted 2019-11-08 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-12

CONDITIONS: Lymphoma, B-Cell
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non-intervention — non-interventional, prospective cohort study

SUMMARY:
Central nervous system lymphoma (CNSL) is a rare brain tumor constituting 3% of all newly diagnosed brain tumors, and 2% to 3% of all cases of non-Hodgkin lymphoma. There are two subtypes of CNSL. Owing to its low incidence, there is limited prospective and/or randomized data to guide the therapy of CNSL. Current knowledge about optimal diagnostic, prognostic and therapeutic strategies of CNSL is urged.

The immune system plays a fundamental role in controlling and eradicating cancer but is held in check by inhibitory receptors and ligands. These immune checkpoint pathways, which normally maintain self-tolerance and limit collateral tissue damage during anti-microbial immune responses, can be co-opted by cancer to evade immune destruction. A plethora of regulatory molecules have been identified. Among them, three have been studied most intensively: cytotoxic T lymphocyte antigen 4 (CTLA4) binding to CD80 or CD86, programmed cell death protein 1 (PD-1) binding to PD-1 ligand 1 (PD-L1) or PD-L2, and SIRPαbinding to CD47. Agents inhibiting CTLA-4, PD1, PD-L1 and CD47 are showing compelling antitumor activity in several solid and hematological cancers. Exploring the role of immune checkpoint pathways in CNSL may help us to establish the rational targeted therapies.

In this study, the investigators will investigate the protein expression of several specific molecules in immune checkpoint pathways such as PD-L1, PD-L2 and CD47 in the large neurological resection specimens by immunohistochemical staining of patients with CNSL. Besides, the concentrations of above molecules and other prognostic relevant factors such as chemokine CXCL13, Interleukin-10 and soluble CD19 in the cerebrospinal fluid (CSF) at initial diagnosis and after treatment will be evaluated using enzyme-linked immunosorbent assays. About 100 patients with CNSL will be recruited. The protein expression of the above molecules will be correlated with the clinical outcome of patients with CNSL. The feasibility of adopting these CSF molecules as useful diagnostic or prognostic biomarkers in CNSL will also be investigated.

DETAILED DESCRIPTION:
Goal The goal and purpose of this study is to investigate the clinical implications and functional roles of immune checkpoint pathways in CNSL.

There are two specific aims:

1. The adoption of protein expression of immune checkpoint pathways (CTLA-4, PD-L1, PD-L2, CD47) as a prognostic factor in patients with PCNSL. To fulfill this aim, the protein expression of CTLA-4, PD-L1, PD-L2, and CD47 in the neurosurgical resection specimens of patients with PCNSL will be evaluated by immunohistochemistry (IHC) techniques. The results will be correlated with clinical features and outcome of the patients with CNSL. Once parameters for these tissues are established it will be possible to speculate about the tumor grade, survival and response to treatment of these patients.
2. The feasibility of adopting CSF CTLA-4, PD-L1, PD-L2, and sCD47 as useful diagnostic and prognostic biomarkers in patients with CNSL. To fulfill this aim, the concentrations of CSF CTLA-4, PD-L1, PD-L2 and sCD47 will be evaluated at the timings of initial diagnosis and after each cycle of systemic chemotherapy by enzyme-linked immunosorbent assays (ELISAs). The concentrations of these CSF molecules at initial diagnosis will be correlated with the prognosis of patients with CNSL. Besides, the investigators will compare the serial follow-up concentrations of these markers after each cycle of systemic chemotherapy to find out whether the presence of decreased concentrations will response to therapy.

This may help to discovery new diagnostic, prognostic and potential therapeutic strategies for patients with CNSL.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with newly diagnosed PCNSL at National Taiwan University Hospital from January 1996 to December 2020
* 2. Patients aged 20 years and older

Exclusion Criteria:

* 1. Subjects who are involved in any interventional treatment that might change experimental biomarkers, such as PD-L1 inhibitor, PD-1 inhibitor, anti CTLA-4 agents…etc before tumor and CSF sampling.
* 2. Pregnancy or breast-feeding

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed PCNSL at National Taiwan University Hospital from January 1996 to December 2020
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2016-10-27 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | 5 years
  OS was measured from the date of the first diagnosis to the end of the follow-up period, death from any cause, or the date of the last known follow-up examination.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 5 years
  PFS was measured from the date of the first diagnosis until the end of the follow-up period, the date of relapse or progressive disease, death from any cause, or the last known follow-up examination, whichever came first.
Treatment response | 1 year
  Tumor responses were assessed through brain MRI or CT in all patients after two or three cycles of chemotherapy as well as at treatment completion.

CONTACTS AND LOCATIONS:
Overall Officials: Chieh-Lung Cheng, Dr, Principal Investigator — NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No